CLINICAL TRIAL: NCT02181205
Title: Sphenopalatine Ganglion Block for Treatment of Postdural Puncture Headache: A Prospective Randomized Double Blind Placebo Controlled Study
Brief Title: Sphenopalatine Ganglion Block for Post-Dural Puncture Headache
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no eligible participant , technical difficulty, feasiblity
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-024
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-02

CONDITIONS: Postdural Puncture Headache; Sphenopalatine Ganglion Block
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Experimental): sphenopalatine ganglion block performed with normal saline as the placebo
  Interventions: Drug: placebo
- bupivacaine (Active Comparator): sphenopalatine ganglion block performed with bupivacaine
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: bupivacaine
  Arms: bupivacaine
Drug: placebo
  Arms: placebo

SUMMARY:
The investigators are attempting to determine a less invasive method of treatment for postdural puncture headaches that can occur after regional anesthesia. The investigators will be evaluating the relief of headache with those subjects receiving treatment with a sphenopalatine ganglion block with bupivacaine versus placebo, evaluating the incidence of epidural blood patch, pain score of headache at 1 hour, then 24, 48, and 72 hours lower with post study treatment versus placebo, and potential side effects of those patients receiving study therapy as well as epidural blood patch.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists assigned class I-III
* age >/= 18 years
* experiencing a postdural puncture headache within 7 days of neuraxial analgesia rated >3/10 pain score

Exclusion Criteria:

* allergy to study medications <18 years of age pain score on presentation </=3/10 for headache

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12-31 (Estimated); Study Completion 2016-12-31 (Estimated)

PRIMARY OUTCOMES:
verbal pain score | 1 hour
  a reduction in headache verbal pain score by 3

SECONDARY OUTCOMES:
epidural blood patch | 7 days
  evaluating the decrease in the necessity of an epidural blood patch to treat the postdural puncture headache
patient satisfaction | 1 hour
  patient satisfaction with headache pain relief at 1 hour post treatment
pain score | 30 minutes
  verbal pain score 30 minutes post study treatment
pain score | 7 days
  verbal pain score 7 days post study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Pan, MD, MSEE, Principal Investigator — Wake Forest School of Medicine-Anesthesiology
Locations (1):
- Novant Health Forsyth Medical Center, Winston-Salem, North Carolina, United States